CLINICAL TRIAL: NCT02234024
Title: Oral Supplementation of Gangliosides - A Potential Treatment for GM3 Synthase Deficiency
Brief Title: Oral Supplementation of Gangliosides to Treat a Rare Metabolic Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: DDC Clinic - Center for Special Needs Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDC-62314
Record Dates: First submitted 2014-09-03; First posted 2014-09-09 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: GM3 Synthase Deficiency
MeSH Terms: conditions — Amish Infantile Epilepsy Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supplementation of gangliosides (Experimental): Supplementation of dairy-derived concentrated gangliosides
  Interventions: Dietary Supplement: Supplementation of dairy-derived concentrated gangliosides.

INTERVENTIONS:
Dietary Supplement: Supplementation of dairy-derived concentrated gangliosides.

SUMMARY:
The purpose of this pilot project is to see if a supplemental form of dietary gangliosides can serve as a potential treatment for the rare metabolic condition called ganglioside GM3 synthase deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of GM3 synthase deficiency

Exclusion Criteria:

-

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Body length compared to normal pediatric growth curves. | Quarterly measures- change from baseline over 24 months.
Change in scores of standardized developmental assessments (Vineland & Batelle) | Quarterly measures - change from baseline over 24 months
Body Weight compared to normal pediatric growth curves | Quarterly measurements from baseline over 24 months
Head circumference compared to normal pediatric growth curves. | Quarterly measures from baseline over 24 months

SECONDARY OUTCOMES:
Concentration of ganglioside GM3 in blood plasma | Six times per year over 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Heng Wang, MD PhD, Principal Investigator — DDC Clinic